CLINICAL TRIAL: NCT00574860
Title: A Phase 3, Multi-center, Randomized, Double-Blind, Placebo- Controlled Study to Assess the Efficacy and Safety of EN3285 for the Prevention or Delay to Onset of Severe Oral Mucositis in Patients With Head and Neck Cancer Receiving Chemoradiotherapy
Brief Title: EN3285 for the Prevention or Delay of Oral Mucositis in Patients With Head and Neck Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Additional research
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EN3285-301
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Oral Mucositis; Head and Neck Cancer
Keywords: Oral Mucositis; Chemoradiation therapy; Head and neck cancer
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EN3285 (NAC ProGelz) (Experimental): The EN3285 arm is the product under development
  Interventions: Drug: EN3285
- No active ingredients (placebo) (Placebo Comparator): This will be an oral product that contains no active ingredient
  Interventions: Drug: Placebo
- Standard of Care (Other): This arm will reflect the typical standard of care for the patient
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: EN3285 — Oral rinse
  Arms: EN3285 (NAC ProGelz)
Drug: Placebo — Oral rinse
  Arms: No active ingredients (placebo)
Other: Standard of care — This will be the therapy most commonly used the the institution treating the patient
  Arms: Standard of Care

SUMMARY:
Randomized, double-blind, placebo-controlled study for the treatment of head and neck cancer(HNC), to assess the ability of EN3285 to prevent or delay the onset of severe oral mucositis(OM).

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled study will be conducted in patients receiving chemoradiotherapy (ChemoRT) for the treatment of head and neck cancer(HNC), to assess the ability of EN3285 to prevent or delay the onset of severe oral mucositis(OM). The study includes a treatment period of up to 8 weeks, based on the patients' prescribed treatment plan, with a follow-up period of 12 months following completion of radiotherapy (RT).

ELIGIBILITY:
Significant Inclusion Criteria:

* 18 years and older
* newly diagnosed SCC of the oral cavity and/or oropharynx, and are intended for treatment with ChemoRT.
* Have a clinical plan to receive a minimum of 60 Gy to the oral cavity and/or oropharynx
* Chemotherapy: cisplatin
* Have a WBC ≥3500 per cubic millimeter
* Have a platelet count ≥100,000 per cubic millimeter
* Have adequate renal function as determined by the principal investigator prior to enrollment
* Are willing and able to undergo oral assessments
* Have a Karnofsky Performance Status score ≥70

Significant Exclusion Criteria:

* Have OM or other oral conditions at study entry
* Plan to use Amifostine, Pilocarpine, Cevimeline or Bethanechol
* Are using a pre-existing feeding tube for nutritional support at study entry
* Plan to use any drug for the treatment or prevention of OM
* Have had any prior radiotherapy to the head and neck
* Have had prior chemotherapy within 6 months preceding enrollment
* Plan to have concurrent chemotherapy, other than those regimens specified under inclusioncriteria
* Have received other investigational drugs in the 30 days preceding initiation of study drug or during administration of study drug
* Have medical conditions that require the use of chronic steroid therapy
* Have the inability to undergo repeat treatments,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
NCI v3 to measure severity of OM | At 50 Gy

SECONDARY OUTCOMES:
WHO criteria for measuring severity of OM | At 50 Gy

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chambers, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Commonwealth ENT, Louisville, Kentucky
  - MD Anderson Cancer Center, Houston, Texas